CLINICAL TRIAL: NCT05372133
Title: PROSPR: PeriopeRative Opioid Stewardship Program of Research (Phase 4 Split Script Study)
Brief Title: Split Scripts for Pediatric Supracondylar Fracture Repairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Conor McDonnell, Principal Investigator, Associate Professor, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000079222
Record Dates: First submitted 2022-02-15; First posted 2022-05-12 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Analgesics, Opioid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Split Script (Experimental): Participants will receive four doses initially, with opportunity to obtain four additional doses if required
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Children will be provided with morphine for at-home pain management following supracondylar fracture repair
  Other Names: Opioid

SUMMARY:
This study is designed to test the hypothesis that increased electronic order-set compliance and focused education will decrease the amount of unconsumed opioid entering and remaining in the home after pediatric supracondylar fracture repair

The proposed study will address the hypothesis with the following objectives:

1. investigators will increase compliance with previously implemented standardized precision-based electronic discharge order sets;
2. investigators will introduce part-fill opioid prescriptions for supracondylar fracture repairs;
3. investigators will increase parental compliance with home administration of simple (non-opioid) analgesics;
4. investigators will decrease opioid amount remaining in the home pre and post 3-week follow up.

DETAILED DESCRIPTION:
Canada has one of the highest opioid prescribing rates in the world (United Nations, 2018). In 2017, Health Quality Ontario published a major report that identified the number of opioid prescriptions following surgery were second only to those following dentist office visits. As a result, Health Quality Ontario made the reduction of opioid prescribing ('Cut the Count)' their number one provincial healthcare priority of 2019.

To date, investigators have decreased MME amount of opioid entering the home post-supracondylar fracture repair at approximately 10 MME per patient and increased the rate of return of unused drug by 10 MME per patient. The Hospital for Sick Children alone performs some 200 such surgeries per year, representing 4,000 mg of morphine (four grams) that the community is no longer exposed to. This is only one surgery type in one hospital; expansion of our methodology to other surgeries (currently expanding to dental and cleft palates) and other institutions will dramatically decrease unintentional but iatrogenic home exposure of children and families to unwarranted and dangerous drugs.

This latest study aims to address all three steps outlined in the 2020-2021 Health Quality Ontario surgical mandate for children discharged from The Hospital for Sick Children after supracondylar fracture repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type II or Type III supracondylar fractures undergoing surgical wire placement or pinning that return to fracture clinic at three weeks for removal of pins/wires.

Exclusion Criteria:

* Patients who are not prescribed morphine following a supracondylar fracture repair surgery

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Amount of morphine milligram equivalents (MME) used at home per SCF patient between July 2022 and October 2023 | 3 days following discharge from hospital
  Recording of how much morphine (mgs or doses) was used at home following supracondylar fracture repair surgery

SECONDARY OUTCOMES:
Compliance with orders for home use of acetaminophen and ibuprofen per SCF patient between July 2022 and October 2023 | 3 days following discharge from hospital
  Recording of whether Tylenol and Advil were used at-home following supracondylar fracture repair surgery
Amount of morphine milligram equivalents (MME) returned to pharmacy per SCF patient between July 2022 and October 2023 | 3 weeks following discharge (aligns with pin/wire removal at fracture clinic)
  Recording of how much morphine was returned to the hospital pharmacy
Healthcare provider compliance to discharge order set | Up to 100 weeks
  Recording of how often healthcare providers deviate from the standardized electronic discharge order set

CONTACTS AND LOCATIONS:
Overall Officials: Conor Mc Donnell, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No